CLINICAL TRIAL: NCT04280978
Title: Pragmatic Abilities in Children With Acquired Brain Injury: Assessment and Analysis With the ABaCo Test
Brief Title: Pragmatic Abilities in Children With Acquired Brain Injury
Acronym: ABIabc
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 01.2020 Oss.
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Acquired Brain Injury; Pragmatic Communication Disorder
MeSH Terms: conditions — Brain Injuries; Social Communication Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aquired Brain Injury: Suitable potential participants would be children with ABI, at least 6 months post onset, from 6 to 11 years old, without diagnosis of aphasia, dysarthria, apraxia, and/or sensorial difficulties (visual and hearing), with Italian as a first language.
  Interventions: Diagnostic Test: ABI ABC

INTERVENTIONS:
Diagnostic Test: ABI ABC — The assessor will administer ABaCo test through a computer device and she will marked the responses on a paper sheet. Video recordings are needed only to allow an impartial scoring. In fact, an external trained judge will do the scoring.
  Furthermore the linguistic abilities will be assessed through the administration of some subtests of the Italian battery "BVL 4-12". In particular, the researcher will administer the following subtests: "naming", "lexical comprehension" and "grammatical comprehension".
  Moreover, some neuropsychological abilities will be analysed using the test "BVN 5-11". In addition, the theory of mind and the non-verbal IQ will be assessed.
  The Socio-Economic-Status of the family involved in the research will also be investigated, considering its importance on the rehabilitation outcomes.
  Other Names: ABaCo test

SUMMARY:
Although neuroplasticity of the brain is high in childhood, some neuropsychological sequelae could persist over the long term in children with Acquired Brain Injury (ABI). Many children with TBI, show deficits in pragmatic abilities that usually persist. Pragmatic difficulties have been observed also in children with sequelae of brain neoplasms .

The lack of validated assessment tools for this population is described in literature. This limit is also valid for the tests that assess pragmatic abilities. The tests that SLPs usually administer investigate only the comprehension of verbal pragmatic and, sometimes the comprehension of linguistic and emotional prosody as well. This could lead to the risk that, sometimes, some pragmatic abilities might not be included in the evaluation. Moreover, it leads to a harder definition of the treatment aims and a harder objective demonstration of treatment outcomes.

For these reasons, it is important to use an assessment tool that provides information on all the pragmatic abilities, not only in input but also in output. Some Italian researchers, recently, developed a test that investigates all these areas. It is called "ABaCo", and it is based on the Cognitive Pragmatics Theory. This theory is focused on cognitive processes underlying human communication.

This test is standardized on a normative group of 300 adults. It was developed with the aim of assessing pragmatic abilities in adults with brain injuries. The assessor shows short videos to the patient, and he/her has to complete or understand the interaction transmitted through different communication channels. The authors also created an adaptation of this test for children aged 5 to 8.6 years old, modifying some items. After that, they administered this adaptation of the test to 390 healthy children. In another study, the authors administered this version of the batteries to children with autism spectrum disorders and to a control group of healthy children, matched by age and sex.

Considering all the studies that already exist for the application of this assessment tool in childhood and adolescence, and the perspective of a standardization for developmental ages, this study aims to investigate whether this test could be useful to detect pragmatic difficulties also in children with ABI.

DETAILED DESCRIPTION:
This project involved two different experimental populations: children with Acquired Brain Injury. Moreover, it includes a wider investigation; in fact, it involves the assessment, not only of linguistic and pragmatic abilities but also of neuropsychological abilities and the theory of mind.

Approximately 30 children with Acquired Brain Injury will be involved in the study.

The data will be collected through the administration of the adapted version of ABaCo test, individually, to each subject involved in the study. The assessment will be conducted in the IRCCS Eugenio Medea. The assessor will administer ABaCo test through a computer device and she will marked the responses on a paper sheet. Video recordings are needed only to allow an impartial scoring. In fact, an external trained judge will do the scoring. The researchers will complete the scoring process within two weeks from the acquisition of the recordings, after that they will destroy the videos.

Furthermore the linguistic abilities will be assessed through the administration of some subtests of the Italian battery "BVL 4-12". In particular, the researcher will administer the following subtests: "naming", "lexical comprehension" and "grammatical comprehension".

Moreover, some neuropsychological abilities will be analysed using the test "BVN 5-11". In addition, the theory of mind and the non-verbal IQ will be assessed.

The Socio-Economic-Status of the family involved in the research will also be investigated, considering its importance on the rehabilitation outcomes , using a questionnaire realized, based on the "Four Factor Index of Social Status".

ELIGIBILITY:
Inclusion Criteria:

* italian
* 6 to 11 years old
* at least 6 months after ABI onset

Exclusion Criteria:

* diagnosis of aphasia, dysarthria, apraxia, and/or sensorial difficulties (visual and hearing)

Ages: 6 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: Acquired Brain Injury
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-06 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
ABaCo | 3 years after ABI
  ABaCo test

SECONDARY OUTCOMES:
BVL 4-12 | 3 years after ABI
  Italian neuropsychological test "BVL 4-12"
BVN 5-11 | 3 years after ABI
  Italian neuropsychological test "BVN 5-11"
QI | 3 years after ABI
  non-verbal Intelligence Quotient

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No